CLINICAL TRIAL: NCT05962099
Title: Defining Circadian Metabolism in Non-alcoholic Fatty Liver Disease
Acronym: DECIMAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 15296
Record Dates: First submitted 2023-05-22; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-05

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adipose and skeletal muscle tissue, urine, serum/plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD
  Interventions: Behavioral: Lifestyle and weight loss advice
- Controls (non-NAFLD)

INTERVENTIONS:
Behavioral: Lifestyle and weight loss advice — Commercially available lifestyle and weight loss intervention
  Groups: NAFLD

SUMMARY:
The investigators will conduct an open label, experimental medicine study exploring the diurnal patterns of hepatic lipid metabolism in NAFLD and non-NAFLD participants (determined by Transient elastography (TE) with controlled attenuation parameter (CAP)). We will also determine whether the diurnal patterns of lipid metabolism in NAFLD participants can be modified using lifestyle and weight loss intervention. Fourteen participants without NAFLD will have morning and evening metabolic investigations (visit 1M & 1E) to assess for changes in lipid flux pathways across the course of the day. After morning and evening investigations their involvement in the clinical study will then end. Seventeen NAFLD participants will also have identical baseline morning and evening investigation after which they will be enrolled into a 12-week lifestyle and weight loss programme. After 12-weeks, all 17 participants with NAFLD will have a follow up CAP, and morning and evening metabolic investigations (visit 2M & 2E).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* BMI 25-50 kg/m2
* Age 18-75 years

Exclusion Criteria:

* A diagnosis of type 1 diabetes
* Type 2 diabetes controlled with medications other than metformin (within last 3 months)
* Shift working patterns in last 3-months or if likely to work shifts during study period.
* Current or recent (<3-months) use of weight loss medications
* Current or recent use of oral contraceptive pill or hormone replacement therapy (within last 3-months)
* Pregnancy
* A blood haemoglobin <120mg/dL
* History of alcoholism or a greater than recommended alcohol intake (Recommendations > 21 units on average per week for men and > 14 units on average per week for women)
* Haemorrhagic disorders
* Treatment with anticoagulant agents
* Other co-morbidities that in the eyes of the investigators may affect data collection
* Any medical condition in the opinion of the investigator that might impact upon safety or validity of the results
* Transient elastography (TE) controlled attenuation parameter (CAP) of between 216-305 dB/m

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NAFLD participants Confirmed by transient elastography (TE) with controlled attenuation parameter (CAP) ≥306 dB/m
  Non-NAFLD Confirmed by transient elastography (TE) with controlled attenuation parameter (CAP) ≤215 dB/m
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in hepatic fatty acid synthesis as measured by incorporation of 2H2 palmitate from 2H2O into very low density lipoprotein triglyceride (VLDL-TG) between morning and evening | 12 hours

SECONDARY OUTCOMES:
Difference in morning and evening glucose production and disposal (of a labelled stable isotope tracer) during a two-step hyperinsulinaemic-euglycaemic clamp | 12 hours
Difference in morning and evening glucose oxidation measured by incorporation of 13C in breath CO2 across a 2-step hyperinsulinemia euglycaemic clamp | 12 hours
Changes in diurnal patterns of hepatic fatty acid synthesis after weight loss programme (measured by incorporation of 2H2 palmitate from 2H2O into very low density lipoprotein triglyceride (VLDL-TG) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No